CLINICAL TRIAL: NCT03175445
Title: Sexual Dimorphism Analysis in Egyptian Population by Locating the Mandibular Canal Using Cone-beam Computed Tomography: an Observational Cross Sectional Study
Brief Title: Sexual Dimorphism Analysis in Egyptian Population by Locating the Mandibular Canal Using CBCT
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Arwa Mousa, assistant lecturer of oral radiology d, Cairo University
Other Study IDs: CEBD-CU-2017-05-09
Record Dates: First submitted 2017-05-30; First posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Gender Identity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- mandible CBCT scans in males: 74 males CBCT scan by planmeca promax 3D Mid machine using 90 kVp, 10 mA, 14 seconds and 200×60 mm FOV with a 0.2 mm voxel size.
  Interventions: Other: CBCT scan by planmeca promax
- mandible CBCT scans in female: 74 females CBCT scan by planmeca promax 3D Mid machine using 90 kVp, 10 mA, 14 seconds and 200×60 mm FOV with a 0.2 mm voxel size
  Interventions: Other: CBCT scan by planmeca promax

INTERVENTIONS:
Other: CBCT scan by planmeca promax — software measurement tool of CBCT

SUMMARY:
Sexual dimorphism analysis in Egyptian population by locating the mandibular canal using cone-beam computed tomography: an observational cross sectional study

DETAILED DESCRIPTION:
Many studies from different countries such as United States, China, Japan, and Europe were done to observe the distinct morphologic and morphometric manifestations of sexual dimorphism. Accordingly, it is mandatory to target a specific population with their unique skeletal features.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above.
* Absence of large pathological lesions in mandible.
* Dentulous patients

Exclusion Criteria:

* Patients younger than 18 years old
* Presence of large pathological lesions in mandible
* Completely edentulous patients.

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult Egyptian population
Sampling Method: Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2017-12-30 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Anterior ramus width , posterior ramus width | 2 years
  distance from mandibular foramen to most anterior and posterior points of ramus respectively

CONTACTS AND LOCATIONS:
Overall Officials: Arwa Mousa, Principal Investigator — Cairo University
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided